CLINICAL TRIAL: NCT01591447
Title: An Open-Label Study to Evaluate the Efficacy and Safety of a Single-Dose of Oral CEM-101 in the Treatment of Male and Female Patients With Uncomplicated Urogenital Gonorrhea
Brief Title: Safety and Efficacy Study of Single-Dose Oral CEM-101 in Patients With Uncomplicated Urogenital Gonorrhea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE01-202
Record Dates: First submitted 2012-05-02; First posted 2012-05-04 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Uncomplicated Urogenital Gonorrhea
MeSH Terms: interventions — solithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Solithromycin (CEM-101) (Experimental): A single oral dose of 1200 mg solithromycin
  Interventions: Drug: solithromycin
- Solithromycin 1000 mg (Experimental): A single oral dose of 1000 mg solithromycin
  Interventions: Drug: Solithromycin (CEM-101)

INTERVENTIONS:
Drug: solithromycin — A single oral dose of 1200 mg solithromycin (CEM-101)
  Arms: Solithromycin (CEM-101)
Drug: Solithromycin (CEM-101) — A single oral dose of 1000 mg solithromycin
  Arms: Solithromycin 1000 mg

SUMMARY:
To determine the safety and efficacy of a single dose of solithromycin (CEM-101) for the treatment of uncomplicated urogenital gonorrhea.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a urogenital gonococcal infection (prior culture, NAAT test, Gram stain, sexual contact)
2. Willing to abstain from anal, oral, or vaginal sexual intercourse or use condoms until study completion.
3. Females of childbearing potential (including females less than 2 years post-menopausal) must have a negative pregnancy test at enrollment.

Exclusion Criteria:

1. Confirmed, or suspected, complicated or systemic gonococcal infections such as pelvic inflammatory disease, arthritis, or endocarditis.
2. Known HIV, chronic hepatitis B, or hepatitis C infection.
3. Known concomitant infection which would require additional systemic antibiotics.
4. Use of systemic or intravaginal antibiotics within 30 days prior to study drug administration.
5. Current use of corticosteroid drugs or other immunosuppressive therapy.
6. Cytotoxic chemotherapy or radiation therapy within the previous 3 months.
7. Known significant renal, hepatic, or hematologic impairment.
8. History of intolerance or hypersensitivity to macrolide antibiotics.
9. Any concomitant condition that, in the opinion of the Investigator, would preclude an evaluation of a response or make it unlikely that the contemplated course of therapy and follow-up could be completed (e.g., life expectancy <30 days).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The bacterial eradication rate, as measured by conversion from positive Neisseria gonorrhoeae baseline urethral or cervical culture to negative | 3 to 9 days after study drug dosing

SECONDARY OUTCOMES:
Safety and tolerability of a single oral dose of CEM-101 in adult patients with uncomplicated urogenital gonorrhea | One day after study drug dosing, and 3 to 9 days after study drug dosing
  Adverse event reporting, clinical laboratory evaluations
The bacterial eradication of rectal or pharyngeal gonococcal infection (if positive culture at baseline) | 3 to 9 days after study drug dosing
Eradication or persistence of N. gonorrhoeae nucleic acid (as measured by positive NAAT assay) from urethral and cervical specimens | 3 to 9 days after study drug dosing
Eradication or persistence of Chlamydia trachomatis nucleic acid (as measured by positive NAAT assay) from urethral and cervical specimens | 3 to 9 days after study drug dosing
In vitro minimum inhibitory concentrations (MICs) of gonococcal strains isolated | Baseline and (if applicable) 3 to 9 days after study drug dosing

CONTACTS AND LOCATIONS:
Overall Officials: Edward W Hook, MD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - Jefferson County Department of Health, Birmingham, Alabama
  - Harborview STD Clinic, Seattle, Washington

REFERENCES:
- [Derived] Hook EW 3rd, Golden M, Jamieson BD, Dixon PB, Harbison HS, Lowens S, Fernandes P. A Phase 2 Trial of Oral Solithromycin 1200 mg or 1000 mg as Single-Dose Oral Therapy for Uncomplicated Gonorrhea. Clin Infect Dis. 2015 Oct 1;61(7):1043-8. doi: 10.1093/cid/civ478. Epub 2015 Jun 18. PMID 26089222